CLINICAL TRIAL: NCT02030691
Title: Tolerance of Nasal High Frequency Percussive Ventilation Versus Nasal CPAP in Neonatal Respiratory Distress in Term and Preterm (> 33 Weeks of Gestation) Neonates
Brief Title: Tolerance of nHFPV Versus nCPAP in Neonatal Respiratory Distress
Acronym: TONIPEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2013/10
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Neonatal Respiratory Distress
Keywords: Neonatal respiratory distress; nHFPV; nCPAP; cerebral tissue oxygenation; NIRS
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nCPAP - nHFPV (Experimental): Eligible patient received after randomization nCPAP or nHFPV for 15 minutes then after the 15 minutes, they received the seconde non invasive device for 15 minutes. Study end 30 minutes after randomization or before if mechanical ventilation is required.
  Interventions: Device: Nasal continuous airway positive pressure (nCPAP); Device: Nasal high frequency percussive ventilation (nHFPV)
- nHFPV - nCPAP (Experimental): Eligible patient received after randomization nCPAP or nHFPV for 15 minutes then after the 15 minutes, they received the seconde non invasive device for 15 minutes. Study end 30 minutes after randomization or before if mechanical ventilation is required.
  Interventions: Device: Nasal continuous airway positive pressure (nCPAP); Device: Nasal high frequency percussive ventilation (nHFPV)

INTERVENTIONS:
Device: Nasal continuous airway positive pressure (nCPAP)
Device: Nasal high frequency percussive ventilation (nHFPV)

SUMMARY:
Respiratory distress is the main cause of morbimortality in preterm and term neonates. In most of the case, these babies required the use of positive end expiratory pressure (PEEP) delivered by a non invasive device. Nasal continuous airway positive pressure (nCPAP) is widely used in neonatal intensive care unit. Nasal high frequency percussive ventilation (nHFPV) can be used as non invasive device to deliver PEEP, and improved lung clearance.

We hypothesized that nHFPV can be used to deliver PEEP in preterm and term newborn with respiratory distress with the same tolerance as nCPAP. To compare the tolerance of these devices we used cerebral tissue oxygenation (rSO2c) measured by near infrared spectroscopy (NIRS).

DETAILED DESCRIPTION:
The objective is to compare nHFPV versus nCPAP tolerance for providing PEEP in newborn respiratory distress.

High frequency percussive ventilation (HFPV) is a pressure limited, time-cycled, high-frequency mode of ventilation that delivers subphysiologic tidal volumes at rapid rates and that can be used via an endotracheal tube, a nasal probe or a face mask. In burned children, it has been shown to provide the same or improved oxygenation and ventilation at lower peak pressure when compared with conventional ventilation. In neonates, HFPV has been described in hyaline membrane disease and acute respiratory failure ventilation with improvement in oxygenation, significant decrease in PaCO2 and no change in central hemodynamics and we recently shown that nasal HFPV is more effective than nasal continuous positive airway pressure in transient tachypnea of the newborn. This stud is a cross-over clinical trial. For each patient enrolled, the 2 respiratory devices (nHFPV and nCPAP) were used one after the other for 15 minutes each. Randomization determines which device to use in first (group A nCPAP then nHFPV, group B (nHFPV then nCPAP). During the experiment, rSO2c is continuously recorded by NIRS, and oxygenation and capnia are monitored in a non invasive way by transcutaneous oxygen saturation and transcutaneous capnia measurement. Ventilators' setting (PEEP, FiO2) will be modified to achieve oxygen and capnia targets (SpO2 > 90%, and under 95% if FiO2>0.21, Capnia between 5 to 7 kPa). Duration of patient follow up is 30 minutes. After these 30 minutes, if PEEP is always needed, patients undergo nCPAP. If needed during the experiment, patients can receive mechanical ventilation (the criteria for mechanical ventilation are the same as those used in clinical practice).

ELIGIBILITY:
Inclusion Criteria:

* Inborn neonate.
* Delivered by vaginal delivery or caesarean section.
* Gestational age greater than or equal to 33 weeks of gestation.
* Birth weight > 1kg.
* Respiratory distress with a Silverman score greater than or equal to 4 after 10 minutes of life.
* Signed parental informed consent.

Exclusion Criteria:

* Meconium aspiration syndrome.
* Congenital anomalies such as heart anomalies, congenital cystic adenomatoid malformation, diaphragmatic hernia…

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Measurement of cerebral tissue oxygenation (rSO2c) by near infrared spectroscopy (NIRS). We compared the mean of the variation of rSO2c during the last 5 minutes for each device (nHFPV and nCPAP). | 30 minutes after the inclusion

SECONDARY OUTCOMES:
Measurement of transcutaneous capnia and oxygen saturation; variation of heart rate, breath rate and blood pressure; ventilators' setting (PEEP, FiO2). | 30 minutes after the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Laurent RENESME, MD, Principal Investigator — University Hospital Bordeaux, France; Antoine BENARD, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Service de Néonatalogie - Maternité - Hôpital Pellegrin, Bordeaux, Bordeaux, France